CLINICAL TRIAL: NCT03638947
Title: Reducing Perioperative S. Aureus Transmission Via Use of an Evidence-Based, Multimodal Program Driven by an Innovative Software Platform (OR Path Trac)
Brief Title: Reducing Perioperative S. Aureus Transmission
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intermediate analysis produced strong enough results that full study not needed.
Sponsor: Randy Loftus (Other)
Collaborators: RDB Bioinformatics (Industry)
Responsible Party: Sponsor-Investigator, Randy Loftus, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201802843
Record Dates: First submitted 2018-08-15; First posted 2018-08-20 (Actual); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Staphylococcus Aureus; Health Care Associated Infection; Health Care Worker Patient Transmission
MeSH Terms: conditions — Staphylococcal Infections; Cross Infection

STUDY DESIGN:
Who Masked: Participant
Masking Description: After the patient has signed consent, they will receive a pre-surgical kit that will include swabs to be used in the nares, arm pit and groin area (standard of care). In a 1:1 randomization scheme, one half of the patients will receive povidone-iodine swab in addition to the kit (treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Patient will receive by mail a kit containing swab for the nares, armpit and groin.
- Swab kit plus povidone-iodine soap (Active Comparator): Patient will receive by mail a kit containing swab for the nares, armpit and groin. In addition the patient will receive decolonization treatment including povidone-iodine soap for presurgical cleansing two days prior to surgery.
  Interventions: Device: Swab and decolonization using povidone-iodine cleansing

INTERVENTIONS:
Device: Swab and decolonization using povidone-iodine cleansing — Patient in this group will receive improved environmental cleaning and undergo surveillance using swabs and decolonization cleansing.
  Arms: Swab kit plus povidone-iodine soap

SUMMARY:
The purpose of this study is to prevent the spread of S. aureus, a dangerous bacterium, within the operating room and between patients undergoing surgery.

DETAILED DESCRIPTION:
The purpose of this study is to prevent the spread of S. aureus, a dangerous bacterium, within the operating room and between patients undergoing surgery. The investigators will combine several approaches in a "bundle" of activities to achieve this goal. The bundle will include removal of bacterial pathogens from patient skin sites before surgery, from provider hands before, during, and after surgery, from environmental surfaces before and after terminal cleaning, and from the injection ports of patient intravenous catheters. The investigators will use a new surveillance system to evaluate how well the bundle, and each component of the bundle, is working. Surveillance will identify S. aureus transmission events, and movement of S. aureus between reservoirs before, during, and after surgery (perioperative). Surveillance will map transmission events to identify actionable steps to improve the bundle. An infection control perioperative team will act on the surveillance reports to proactively address the action items, and to measure the effect of their efforts for the treatment group. The investigators will compare perioperative S. aureus transmission events for patients receiving the bundle to perioperative S. aureus transmission events for patients receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Undergoing surgery (orthopedic total joint, orthopedic spine, Gynecological/Oncology, thoracic, general, hernia, colorectal, open vascular, plastic surgery and open urological)
* Ability to sign informed consent
* Require general or regional anesthesia

Exclusion Criteria:

* Less than 18 years of age
* Inability to sign informed consent
* Procedures not included above
* Not requiring general or regional anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Loftus, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal

REFERENCES:
- [Background] Vogel TR, Dombrovskiy VY, Lowry SF. Impact of infectious complications after elective surgery on hospital readmission and late deaths in the U.S. Medicare population. Surg Infect (Larchmt). 2012 Oct;13(5):307-11. doi: 10.1089/sur.2012.116. Epub 2012 Oct 19. PMID 23082877
- [Background] Koff MD, Brown JR, Marshall EJ, O'Malley AJ, Jensen JT, Heard SO, Longtine K, O'Neill M, Longtine J, Houston D, Robison C, Moulton E, Patel HM, Loftus RW. Frequency of Hand Decontamination of Intraoperative Providers and Reduction of Postoperative Healthcare-Associated Infections: A Randomized Clinical Trial of a Novel Hand Hygiene System. Infect Control Hosp Epidemiol. 2016 Aug;37(8):888-895. doi: 10.1017/ice.2016.106. Epub 2016 Jun 7. PMID 27267310
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] Boucher HW, Talbot GH, Bradley JS, Edwards JE, Gilbert D, Rice LB, Scheld M, Spellberg B, Bartlett J. Bad bugs, no drugs: no ESKAPE! An update from the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jan 1;48(1):1-12. doi: 10.1086/595011. PMID 19035777
- [Background] Loftus RW, Koff MD, Burchman CC, Schwartzman JD, Thorum V, Read ME, Wood TA, Beach ML. Transmission of pathogenic bacterial organisms in the anesthesia work area. Anesthesiology. 2008 Sep;109(3):399-407. doi: 10.1097/ALN.0b013e318182c855. PMID 18719437
- [Background] Loftus RW, Brown JR, Koff MD, Reddy S, Heard SO, Patel HM, Fernandez PG, Beach ML, Corwin HL, Jensen JT, Kispert D, Huysman B, Dodds TM, Ruoff KL, Yeager MP. Multiple reservoirs contribute to intraoperative bacterial transmission. Anesth Analg. 2012 Jun;114(6):1236-48. doi: 10.1213/ANE.0b013e31824970a2. Epub 2012 Mar 30. PMID 22467892
- [Background] Clark C, Taenzer A, Charette K, Whitty M. Decreasing contamination of the anesthesia environment. Am J Infect Control. 2014 Nov;42(11):1223-5. doi: 10.1016/j.ajic.2014.07.016. Epub 2014 Oct 30. PMID 25444268
- [Background] Loftus RW, Dexter F, Robinson ADM. High-risk Staphylococcus aureus transmission in the operating room: A call for widespread improvements in perioperative hand hygiene and patient decolonization practices. Am J Infect Control. 2018 Oct;46(10):1134-1141. doi: 10.1016/j.ajic.2018.04.211. Epub 2018 Jun 12. PMID 29907449
- [Background] Loftus RW, Dexter F, Robinson ADM. Methicillin-resistant Staphylococcus aureus has greater risk of transmission in the operating room than methicillin-sensitive S aureus. Am J Infect Control. 2018 May;46(5):520-525. doi: 10.1016/j.ajic.2017.11.002. Epub 2018 Jan 4. PMID 29307750
- [Background] Hadder B, Patel HM, Loftus RW. Dynamics of intraoperative Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter transmission. Am J Infect Control. 2018 May;46(5):526-532. doi: 10.1016/j.ajic.2017.10.018. Epub 2018 Feb 12. PMID 29395508
- [Background] Loftus RW, Muffly MK, Brown JR, Beach ML, Koff MD, Corwin HL, Surgenor SD, Kirkland KB, Yeager MP. Hand contamination of anesthesia providers is an important risk factor for intraoperative bacterial transmission. Anesth Analg. 2011 Jan;112(1):98-105. doi: 10.1213/ANE.0b013e3181e7ce18. Epub 2010 Aug 4. PMID 20686007
- [Derived] Loftus RW, Dexter F, Goodheart MJ, McDonald M, Keech J, Noiseux N, Pugely A, Sharp W, Sharafuddin M, Lawrence WT, Fisher M, McGonagill P, Shanklin J, Skeete D, Tracy C, Erickson B, Granchi T, Evans L, Schmidt E, Godding J, Brenneke R, Persons D, Herber A, Yeager M, Hadder B, Brown JR. The Effect of Improving Basic Preventive Measures in the Perioperative Arena on Staphylococcus aureus Transmission and Surgical Site Infections: A Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e201934. doi: 10.1001/jamanetworkopen.2020.1934. PMID 32219407
- See also: Fact Sheet: Obama Administration Takes Actions to Combat Antibiotic-Resistant Bacteria — https://obamawhitehouse.archives.gov/the-press-office/2014/09/18/fact-sheet-obama-administration-takes-actions-combat-antibiotic-resistan
- See also: Updated Guidelines for Evaluating Public Health Surveillance Systems — https://www.cdc.gov/mmwr/preview/mmwrhtml/rr5013a1.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Swab Kit Plus Povidone-iodine Soap
Started | 130 | 106
Completed | 130 | 106
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Swab Kit Plus Povidone-iodine Soap | Total
Number analyzed (Participants) | 130 | 106 | 236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 88 | 60 | 148
  >=65 years | 42 | 45 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 43 | 155
  Male | 18 | 63 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 130 | 106 | 236

OUTCOME MEASURES:

1. Primary Outcome: Quantitate the Reduction of S. Aureus Tranmission
Description: Compare the number of S. aureus transmission events for patients who receive the standard presurgical preparation verses patients who receive decolonization interventions.
Time Frame: Up to 180 days following surgery
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Standard of Care | Swab Kit Plus Povidone-iodine Soap
Number analyzed (Participants) | 130 | 106
events | 1.25 (2.11) | 0.47 (1.13)

2. Secondary Outcome: Identify the Number of Preoperative Patients Positive for S. Aureus Using Collection Kits
Description: To identify the number of patients in the preoperative setting who test positive for S. aureus.
Time Frame: Preoperative
Measure: Number; unit: number of participants
Arm/Group | Standard of Care | Swab Kit Plus Povidone-iodine Soap
Number analyzed (Participants) | 130 | 106
number of participants | 18 | 8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Standard of Care | Swab Kit Plus Povidone-iodine Soap
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/106
Other Adverse Events (participants affected / at risk) | 0/130 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT03638947/Prot_003.pdf
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT03638947/SAP_004.pdf
  • Informed Consent Form (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03638947/ICF_002.pdf